CLINICAL TRIAL: NCT01414933
Title: High Throughput Technologies to Drive Breast Cancer Patients to Specific Phase I/II Trials of Targeted Agents
Acronym: SAFIR-01
Status: Completed | Type: Observational
Sponsor: UNICANCER (Other)
Collaborators: Ministry of Health, France (Other Government); Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Other Study IDs: GRT01/0710 SAFIR-01
Record Dates: First submitted 2011-06-17; First posted 2011-08-11 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Metastasis biopsy and DNA from biopsy
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Biopsy — Breast metastases biopsy

SUMMARY:
High sensitivity to targeted agents has been observed in patients whose tumor cells present a genetic/genomic deregulation of the target (Kit mutation, ERBB2 amplification, EGFR mutations) together with addiction to the given target. More recently, activation of "alternative pathways" (Kras mutation, PI3K mutations) have been reported as a common resistance mechanism to single agent tyrosine kinase inhibitors (trastuzumab, cetuximab).

From these data has emerged the hypothesis that identification of the deregulated pathway through new molecular tools could allow to propose a more tailored targeted regimen.

Based on these concepts, numbers of phase I/II trials enrich their populations in patients presenting specific molecular alterations.

High throughput technologies (array CGH, sequencing, gene expression array) identify deregulated genes. In addition, these technologies determine whether such genomic alterations are single (expected efficacy of single agent) or multiple (rationale for combination). In a pilot study that included 135 patients, we recently performed a combination of array CGH and hot spot mutation array in order to drive patients into phase I/II clinical trials. This study led to the conclusions that high throughput technologies i. are feasible (80%) and robust, ii. identify "targetable" genomic alterations in around 40% of samples.

In the present study, the investigators will perform high throughput technologies to drive 400 metastatic breast cancer patients into specific phase I/II trials.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women with histologically diagnosed breast cancer
* Metastatic relapse or stage IV breast cancer at diagnosis
* Metastases amenable to biopsy
* Age <70 years old
* PS 0/1
* No restriction regarding the number of previous chemotherapy or endocrine therapies

Exclusion Criteria:

* Age <18
* Life expectancy <3 months
* Symptomatic or progressing brain metastases
* Progressive patients at the time of biopsy
* LVEF <50% (MUGA or ultrasonography)
* Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:
* Absolute neutrophil count < 1.5 x 109/L
* Platelet count < 100 x 109/L
* Haemoglobin < 90 g/L
* ASAT/ALAT > 2.5 times the upper limit of normal (ULN) if no demonstrable liver metastases or > 5 times ULN in the presence of liver metastases
* Total bilirubin > 1.5 times ULN
* Creatinine >1.5 times ULN
* Corrected calcium > ULN
* Phosphate > ULN
* Abnormal blood coagulation that contra-indicates biopsy
* Patients deprived of liberty or placed under the authority of a tutor

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women or men with metastatic breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 423 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
number of patients included in early phase trials evaluating targeted drugs | one year after obtaining the molecular profile
  To use whole genome / integrated biology approach to drive patients in early clinical trials. The goal is to include at least 30% of the patients in a clinical trial evaluating targeted agent, according to the molecular alteration detected on high throughput technologies

SECONDARY OUTCOMES:
overall survival | 3 years after inclusion in SAFIR
  To evaluate the efficacy of such patient selection in terms of survival
Progression free survival | 3 years after inclusion in SAFIR
  To evaluate the efficacy of such patient selection in terms of progression free survival
To evaluate the efficacy of such patient selection in terms of survival response rate | 3 years after inclusion in SAFIR
  To evaluate the efficacy of such patient selection in terms of best response rate

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice André, MD phD, Principal Investigator — Institut Gustave Roussy, Villejuif, France
Locations (18):
- France (18):
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Centre Val D'Aurelle, Montpellier
  - Centre Alexis Vautrin, Nancy
  - Institut de Cancérologie de l'Ouest/ René Gauducheau, Nantes
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Institut Jean Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut Curie/ René Huguenin, Saint-Cloud
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] Andre F, Delaloge S, Soria JC. Biology-driven phase II trials: what is the optimal model for molecular selection? J Clin Oncol. 2011 Apr 1;29(10):1236-8. doi: 10.1200/JCO.2010.31.6877. Epub 2011 Feb 22. No abstract available. PMID 21343554
- [Derived] Andre F, Bachelot T, Commo F, Campone M, Arnedos M, Dieras V, Lacroix-Triki M, Lacroix L, Cohen P, Gentien D, Adelaide J, Dalenc F, Goncalves A, Levy C, Ferrero JM, Bonneterre J, Lefeuvre C, Jimenez M, Filleron T, Bonnefoi H. Comparative genomic hybridisation array and DNA sequencing to direct treatment of metastatic breast cancer: a multicentre, prospective trial (SAFIR01/UNICANCER). Lancet Oncol. 2014 Mar;15(3):267-74. doi: 10.1016/S1470-2045(13)70611-9. Epub 2014 Feb 7. PMID 24508104